CLINICAL TRIAL: NCT03373136
Title: Comparison of the Bleeding Risk Between Cold and Hot Snaring Polypectomy for Small Colorectal Polyp: a Randomized Control Trial
Brief Title: Compare Bleeding Risk Between Cold and Hot Snaring Polypectomy for Small Colorectal Polyp: a Randomized Control Trial
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: National Taiwan University Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 201707022RINB
Record Dates: First submitted 2017-11-29; First posted 2017-12-14 (Actual); Last update posted 2020-10-14 (Actual); Status verified 2020-08

CONDITIONS: Colorectal Polyp

STUDY DESIGN:
Who Masked: Participant
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Cold snaring (Experimental): Polypectomy will be done without electrocautery
  Interventions: Device: Polypectomy
- Hot snaring (Active Comparator): Polypectomy will be performed with electrocautery
  Interventions: Device: Polypectomy

INTERVENTIONS:
Device: Polypectomy — Polypectomy during colonoscopy is considered effective to reduce the incidence and mortality of colorectal cancer

SUMMARY:
In this randomized control trial the investigators aim to compare the bleeding complication between cold snaring and hot snaring polypectomy with a large sample size.

DETAILED DESCRIPTION:
The investigators will enroll subjects who receive screening or surveillance colonoscopy with small colorectal polyp, 4 to10 mm in size, from multiple centers in Taiwan. Subjects who are less than 40 years old and has contraindication will be excluded from this study. All the candidates for enrollment will sign the inform consent at the outpatient clinic. Once the candidate has the target lesion, polyp sized 4 to 10 mm, at colonoscopy will be randomized into either cold snaring or hot snaring polypectomy group. In the group with cold snaring, polypectomy will be done without electrocautery. In the hot snaring group, the polypectomy will be performed with electrocautery. The bowel preparation and colonoscopy insertion are the same in both groups as conventional colonoscopy method. The colonoscopy will be performed by experienced endoscopies who performed more than 100 polypectomies per year.

ELIGIBILITY:
Inclusion Criteria:

* Candidate has the target lesion, polyp sized 4 to 10 mm, at colonoscopy

Exclusion Criteria:

* Subjects who are less than 40 years old and has contraindication will be excluded from this study

Min Age: 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 4270 (Actual)
Dates: Start 2018-02-07 (Actual); Primary Completion 2020-08-14 (Actual); Study Completion 2020-08-30 (Actual)

PRIMARY OUTCOMES:
Delayed bleeding rate | 2 weeks
  Anal bleeding with spontaneously stop; drop of Hb more than 2 gm/dl in comparison with baseline; transfusion needed; hemostasis by : colonoscopy, angiography, surgery

CONTACTS AND LOCATIONS:
Overall Officials: Han-Mo CHIU, M.D., Ph.D., Principal Investigator — Department of Internal Medicine, College of Medicine, National Taiwan University
Locations (1):
- Department of Internal Medicine, College of Medicine, National Taiwan University, Taipei, Taiwan

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Raad D, Tripathi P, Cooper G, Falck-Ytter Y. Role of the cold biopsy technique in diminutive and small colonic polyp removal: a systematic review and meta-analysis. Gastrointest Endosc. 2016 Mar;83(3):508-15. doi: 10.1016/j.gie.2015.10.038. Epub 2015 Nov 9. PMID 26545637
- [Result] Horiuchi A, Nakayama Y, Kajiyama M, Tanaka N, Sano K, Graham DY. Removal of small colorectal polyps in anticoagulated patients: a prospective randomized comparison of cold snare and conventional polypectomy. Gastrointest Endosc. 2014 Mar;79(3):417-23. doi: 10.1016/j.gie.2013.08.040. Epub 2013 Oct 11. PMID 24125514
- [Result] Takeuchi Y, Yamashina T, Matsuura N, Ito T, Fujii M, Nagai K, Matsui F, Akasaka T, Hanaoka N, Higashino K, Iishi H, Ishihara R, Thorlacius H, Uedo N. Feasibility of cold snare polypectomy in Japan: A pilot study. World J Gastrointest Endosc. 2015 Nov 25;7(17):1250-6. doi: 10.4253/wjge.v7.i17.1250. PMID 26634041
- [Derived] Tseng CH, Chang LC, Wu JL, Chang CY, Chen CY, Chen PJ, Shun CT, Hsu WF, Chen YN, Chen CC, Huang TY, Tu CH, Chen MJ, Chou CK, Lee CT, Chen PY, Lin JT, Wu MS, Chiu HM. Bleeding Risk of Cold Versus Hot Snare Polypectomy for Pedunculated Colorectal Polyps Measuring 10 mm or Less: Subgroup Analysis of a Large Randomized Controlled Trial. Am J Gastroenterol. 2024 Nov 1;119(11):2233-2240. doi: 10.14309/ajg.0000000000002847. Epub 2024 May 9. PMID 38775310
- [Derived] Chang LC, Chang CY, Chen CY, Tseng CH, Chen PJ, Shun CT, Hsu WF, Chen YN, Chen CC, Huang TY, Tu CH, Chen MJ, Chou CK, Lee CT, Chen PY, Wu MS, Chiu HM. Cold Versus Hot Snare Polypectomy for Small Colorectal Polyps : A Pragmatic Randomized Controlled Trial. Ann Intern Med. 2023 Mar;176(3):311-319. doi: 10.7326/M22-2189. Epub 2023 Feb 21. PMID 36802753
- [Derived] Chen YN, Chang LC, Chang CY, Chen PJ, Chen CY, Tseng CH, Chiu HM. Comparison of cold and hot snaring polypectomy for small colorectal polyps: study protocol for a randomized controlled trial. Trials. 2018 Jul 6;19(1):361. doi: 10.1186/s13063-018-2743-z. PMID 29980220